CLINICAL TRIAL: NCT05920850
Title: The SHARED Project (Testing a Lung Cancer Screening Intervention for AAM)
Brief Title: The SHARED, Project, Lung Cancer Screening for African American Men (AAM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Rohan Dexter Jeremiah, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-0273
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): 1. A culturally tailored video that provides education about the process of low-dose helical computed tomography (LDCT) lung cancer screening
  2. A culturally tailored shared decision-making tool that educates participants about the shared decision-making process
  3. The use of a flip chart that reinforces the information provided in the video and shared decision-making tool
  4. Navigation support for participants who express interest in LDCT and quitting smoking
  Interventions: Other: Educational Video about LDCT lung cancer screening; Other: A culturally tailored shared decision-making tool; Other: Flip chart; Other: Navigation support

INTERVENTIONS:
Other: Educational Video about LDCT lung cancer screening — A culturally tailored video that provides education about the process LDCT lung cancer screening
Other: A culturally tailored shared decision-making tool — A culturally tailored shared decision-making tool that educates participants about the shared decision-making process
Other: Flip chart — The use of a flip chart that reinforces the information provided in the video and shared decision-making tool
Other: Navigation support — Navigation support for participants who express interest in LDCT and quitting smoking.

SUMMARY:
This study is a single-arm pre-test post-test design with a two-month follow-up assessment. The study aims to provide support to participants in quitting smoking and accessing lung cancer screening through the combination of education interventions and patient navigation (PN)

DETAILED DESCRIPTION:
This study is a single-arm pre-test post-test design with a two-month follow-up assessment. The study aims to provide support to participants in quitting smoking and accessing lung cancer screening through the combination of education interventions and patient navigation (PN). After participant consent the study team will administer a series of surveys to collect the participant's contact information and complete the study's pretest measures. These include a demographic survey, smoking history, lung cancer knowledge, lung screening knowledge, intention to quit/screen, informed to decide, satisfaction survey, and decision conflict survey. The study also consists of three scheduled meetings with the PN lasting up to 60 minutes. The 1st session will be held between 7-14 days after consent. The 2nd session will be held 7-14 after the 1st session and the 3rd session will be held 42-49 days after the 1st session. Additional phone calls will last 10 minutes or less and be focused on specific questions generated by study participants.

In the 1st session the PN will re-orient participant to the goals and objectives of the project and answer participant questions before starting the intervention. The 1st activity will be to show a 3 minute culturally tailored video that will explain the benefits of lung cancer screening for African American Males (AAM) using an internet-enabled device. After completion of the video, the PN will invite the participant to ask any questions that they have and the PN will offer clarifying information. The PN will review with the participant a culturally adapted shared decision-making tool. The participant will complete the posttest surveys as described abov.

In the 2nd session the PN will determine the scheduling and completion of lung cancer screening and Illinois Tobacco Quit Line (ITQL) engagement. The participant will complete the LDCT screening, navigation needs, Quitline Engagement, and decision change surveys

In the 3rd session the PN will determine scheduling, barriers and completion of lung cancer screening and Quitline engagement. The participant will complete LDCT screening check, and a Quitline engagement check

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as African American or Black males
2. Current smokers of any nicotine-containing products
3. Do not self-report a history of lung cancer symptoms
4. Speaks English

Exclusion Criteria:

1. Do not self-identify as African American males
2. Former smokers
3. Self-report a history of lung cancer symptoms
4. Do not speak English

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Assess changes in knowledge, attitudes, risk perception, and intention/ stage of readiness to engage in lung cancer screening and smoking cessation | 1 year
  Number of participants that show an improvement from pretest to posttest
Assess the completion of a healthcare visit for the purpose of lung cancer screening ces | 1 year
  Number of participants that complete lung cancer screening
Assess completion of referral to smoking cessation treatment | 1 year
  Number of participants that completed the referral to smoking cessation treatment to the ITQL

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States